CLINICAL TRIAL: NCT01451333
Title: The EFV Central Nervous System Exposure Sub-study of Encore1: A Randomised, Double-blind, Placebo-controlled, Clinical Trial to Compare the Safety and Efficacy of Reduced Dose Efavirenz (EFV) With Standard Dose EFV Plus Two Nucleotide Reverse Transcriptase Inhibitors (N(t)RTI) in Antiretroviral-naïve HIV-infected Individuals Over 96 Weeks
Brief Title: The Efavirenz (EFV) Central Nervous System Exposure Sub-study of Encore1
Acronym: ENCORE1-CNS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCHECR-ENCORE1-CNS
Record Dates: First submitted 2011-01-05; First posted 2011-10-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infection
Keywords: HIV; Efavirenz; Central Nervous System (CNS); Lumbar puncture; Dose reduction
MeSH Terms: conditions — HIV Infections | interventions — efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced dose Efavirenz arm (Experimental): Patient's on main study that was randomised to receive TDF (300mg qd)/FTC (200mg qd) + EFV (400mg qd; 2 x 200mg + 1 x 200mg placebo qd).
  Interventions: Drug: Efavirenz
- Normal Efavirenz dose arm (Active Comparator): Patient's on main study randomised to receive tenofovir (TDF) (300mg qd)/emtricitabine (FTC) (200mg qd) + EFV (600mg qd; 3 x 200mg qd)
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — 600mg qd; 3 x 200mg qd
  Arms: Normal Efavirenz dose arm
Drug: Efavirenz — 400mg qd; 2 x 200mg
  Arms: Reduced dose Efavirenz arm

SUMMARY:
Persistent HIV infection in the central nervous system (CNS) compartment may put subjects at risk of developing HIV-related brain disease. Important factors associated with the development of HIV-related brain disease include therapeutic concentrations of antiretroviral drugs in the CNS. Conflicting evidence regarding the CNS exposure of the antiretroviral drug used for the encore1 study, efavirenz (EFV) have been described in related studies. There were recent study of two small series assessment of EFV exposure in the cerebral spinal fluid (CSF); one group reported small detectable EFV concentrations, while another observed undetectable EFV exposure in the CSF. Also, in a larger reported series comprising of 80 subjects on EFV-containing antiretroviral therapy, a CSF to plasma concentration suggested that there is limited movement of EFV out of the CSF. In HIV-1 infected subjects at steady state, EFV plasma level parameters are dose proportional following 200mg, 400mg, and 600mg daily doses. The CNS exposure of EFV at different daily dosing has not been described.

ELIGIBILITY:
Inclusion Criteria:

* All subjects entering into the main study protocol at participating centres will be eligible to enter this sub-study.

Exclusion Criteria:

* Existing neurological disease which in the opinion of the investigator would be a contra-indication to lumbar puncture examination
* CNS opportunistic infections in the past 12 weeks of randomisation
* Bacterial or viral meningitis in the past 12 weeks of randomisation
* Head injury requiring medical assessment in the past 12 weeks of randomisation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
comparison of mean CSF concentration of EFV from both doses after week 24. | 24 weeks
  measure the CSF exposure of EFV when dosed at 400mg and 600mg daily. Efavirenz plasma and CSF concentrations will be analysed and CSF:plasma ratios will be compared. Associations between plasma and CSF concentrations and relationship to study clinical parameters will be assessed.

SECONDARY OUTCOMES:
CSF EFV exposure and plasma exposure (CSF:plasma ratio) using statistical analysis | 24 weeks
  The relationship between CSF EFV exposure and plasma exposure (CSF:plasma ratio), both for protein bound and free plasma EFV exposure.
The relationship between CSF EFV exposure and neuropsychiatric side effects using questionnaires and medical assessments | 24 weeks
The relationship between CSF EFV exposure and other study parameters such as race and sex. | 24 weeks
The number of subjects with EFV CSF exposure greater than the postulated CSF IC50 for wild type virus (0.51ng/mL) | 24 weeks
CSF HIV RNA measurement after 12 - 24 weeks of study therapy | 24 weeks
Relationship between plasma HIV RNA and CSF HIV RNA | 24 weeks
CSF biomarker analysis after 12 - 24 weeks of study therapy | 24 weeks
comparison between magnetic resonance (MR) spectroscopy findings and CSF HIV RNA and EFV concentration | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, Dr., Principal Investigator — Imperial College London
Locations (5):
- Medical Group Practice, Berlin, State of Berlin, Germany
- Thailand (2):
  - HIVNAT Research Collaboration, Patumwan, Bangkok
  - Khon Kaen University, Khon Kaen, Changwat Khon Kaen
- United Kingdom (2):
  - Imperial College, St. Mary's Hospital, Clinical Trials Centre, Winston Churchil Wing, London
  - Chelsea and Westminster Hospital, Hiv/gum Laboratory 5th Floor Saint Stephen Centre, London